CLINICAL TRIAL: NCT01420185
Title: Molecular Predictors of Loco-Regional Recurrence in Node Positive Breast Cancer
Brief Title: Identification of Genes That Predict Local Recurrence in Samples From Patients With Breast Cancer Treated on NSABP-B-28
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NSABP B-28 ICSCA; NSABP-B28-ICSC-A
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict whether cancer will come back after treatment.

PURPOSE: This research trial is studying genes that may predict local recurrence in samples from patients with breast cancer. treated on NSABP-B-28

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the association between the 21-gene Recurrence Score and risk of local-regional recurrence (LRR) in node-positive, estrogen receptor- (ER) positive (+) patients treated with cyclophosphamide and doxorubicin hydrochloride (AC) with or without paclitaxel in the NSABP-B-28 trial.
* To evaluate the potential for combining the 21-gene Recurrence Score (RS) with traditional clinico-pathologic factors in order to derive an improved algorithm for prediction of LRR risk and in order to identify subgroups of ER-positive patients with 1-3 or 4 or more positive nodes who do/do not need post mastectomy chest wall radiotherapy (XRT) or regional nodal XRT (irrespective of surgical procedure).
* To evaluate whether the 21-gene RS predicts benefit from adding paclitaxel to AC chemotherapy in reducing risk of LRR, and improving disease-free survival (DFS) and overall survival (OS) in node-positive, ER-positive patients from NSABP-B-28.

OUTLINE: RNA extracted from paraffin-embedded tissue samples are analyzed for gene expression profile by Ribogreen assay and RT-PCR. Results are then compared and analyzed with each patient clinical-pathologic factors, including tumor size, patient age, number of positive nodes (1-3, 4+), tumor grade, and surgery type (mastectomy or lumpectomy).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with breast cancer and enrolled on NSABP-B-28.

  * Estrogen-receptor positive (ER+)
  * Node-positive disease
* Primary tumor tissue samples available
* Treated with cyclophosphamide and doxorubicin hydrochloride and tamoxifen with or without paclitaxel

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stored tissue from participants in protocol NSABP B-28.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Association between low, intermediate, and high 21-gene recurrence score (RS) and risk of LRR | approximately 4 years
Identification of a subgroup of patients who may or may not need radiotherapy after surgery | approximately 4 years
21-gene RS in predicting treatment benefit, reducing LRR risk, and improving DFS and OS in node-positive ER+ patients | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Terry Mamounas, MD, MPH, FACS, Principal Investigator — Aultman Cancer Center at Aultman Hospital

REFERENCES:
- [Derived] Wolmark N, Mamounas EP, Baehner FL, Butler SM, Tang G, Jamshidian F, Sing AP, Shak S, Paik S. Prognostic Impact of the Combination of Recurrence Score and Quantitative Estrogen Receptor Expression (ESR1) on Predicting Late Distant Recurrence Risk in Estrogen Receptor-Positive Breast Cancer After 5 Years of Tamoxifen: Results From NRG Oncology/National Surgical Adjuvant Breast and Bowel Project B-28 and B-14. J Clin Oncol. 2016 Jul 10;34(20):2350-8. doi: 10.1200/JCO.2015.62.6630. Epub 2016 May 23. PMID 27217450